CLINICAL TRIAL: NCT05096585
Title: Sleep Restriction and Altered Sleep Timing on Energy Intake and Energy Expenditure
Brief Title: Sleep Timing on Energy Intake and Energy Expenditure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Jill Kanaley, professor, University of Missouri-Columbia
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: sleep timing 2016786
Record Dates: First submitted 2021-10-14; First posted 2021-10-27 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2023-03

CONDITIONS: Obesity
Keywords: sleep restriction; physical activity; dietary intake; insulin resistance
MeSH Terms: conditions — Obesity; Motor Activity; Insulin Resistance

STUDY DESIGN:
Intervention Model Description: All subjects will complete 3 study conditions with a minimum of one week between each condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- normal sleep (Placebo Comparator): Subjects will go to sleep at their normal bedtime and normal sleep duration (7-9 hr)
  Interventions: Behavioral: Delayed bedtime sleep restriction; Behavioral: Early wake sleep restriction
- delayed bedtime sleep restriction (Experimental): Subjects will go to sleep at 2 hr later than their normal bedtime
  Interventions: Behavioral: Delayed bedtime sleep restriction; Behavioral: Early wake sleep restriction
- early waking sleep restriction (Experimental): Subjects will wake up 2 hr earlier than their normal wake time
  Interventions: Behavioral: Delayed bedtime sleep restriction; Behavioral: Early wake sleep restriction

INTERVENTIONS:
Behavioral: Delayed bedtime sleep restriction — bedtime 2 hr later than their normal bedtime
Behavioral: Early wake sleep restriction — wake time 2 hr earlier than their normal wake time

SUMMARY:
Studies in healthy young adults have shown that abnormal and undesirable physiological changes are a result of chronic sleep curtailment, with implications on inflammatory status, blood glucose regulation, circulating free fatty acids, and insulin sensitivity. Epidemiological studies suggest an increase in energy intake with shortened, sleep and this has been associated with weight gain. Interestingly most studies examining sleep restriction do not consider whether the restricted sleep is due to sleep delay or an advanced wake time. This study will investigate the change in physical activity or food intake during a period of sleep restriction. To date only one study has addressed this question but they only examined one study night and followed their subjects for only 24 hr. The objective of the proposed project is to examine the effects of shortened sleep on potential changes in physical activity and energy intake.

The investigators hypothesize that after several nights of short sleep that different strategies are employed to remain awake and these strategies will also vary whether bed time was delayed or wake time was advanced.

Aim 1: To examine the effects of sleep timing on energy intake and expenditure during periods of sleep restriction

DETAILED DESCRIPTION:
Subjects will have preliminary screening tests. There will be 3 study conditions, with the latter 2 conditions (delayed bed time/advanced wake time) will be completed in a randomized, crossover design. Subjects will wear an activity monitor (actigraph) and sleep monitor (actiwatch) for 6 days. Dietary records and smart phones will be used record energy intake.

For the first experimental condition, the subject will wear the actiwatch and actigraph, and monitor food intake for 6 day of normal sleep. This condition will allow determination of their sleep pattern and when they habitually go to bed (ie. 11 pm - 5 am) and awaken.

On the second condition, the investigators will allow subjects to maintain their usual physical activity and dietary patterns but the investigators will ask subjects to delay the time of going to bed by 2 hr. Subjects will be followed for 4 nights of shortened sleep but data will be collected for 6 days. On the other condition, subjects will go to bed at the usual time but awaken 2 hr earlier that they normally would. Again subjects will monitor their physical activity, hunger/fullness, sleep and energy intake. These latter 2 conditions will be randomized.

Visit 1: Subjects will be provided a verbal explanation of the study and will sign the informed consent if interested. Subjects will then complete questionnaires assessing health history, sleep, morningness and physical activity habits.

Visit 2: Subjects will collect physical activity monitor (actigraph) and sleep monitor (actiwatch) along with surveys to fill out each day about dietary consumption, sleep habits and physical activity, lasting for 6 days. Subjects will also be asked to photograph any food or drink they consume.

Visit 3: Return the actiwatch and actigraph.

Visit 4-5: Repeat of Visit 2-3.

Visit 6-7: Repeat of Visit 2-3.

ELIGIBILITY:
Inclusion Criteria:

Overweight and obese men and women 21-45 years of age BMI of <40 kg/m2 normally active (>5000 steps per day) sleep: 7-9 hours per night

Exclusion Criteria:

type 1 diabetes cardiovascular disease uncontrolled hypertension smoker pregnant recent changes in hormonal birth control night shift workers take regular daytime naps operate heavy equipment Sleep less than 7 hour/night

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
physical activity | 24 hours
  physical activity (percent time in sedentary, light, moderate and vigorous PA)
dietary intake | 24 hours
  macronutrient content (percent carbohydrate, fat and protein intake
physical activity | 24 hours
  Step count (steps/day)
dietary intake | 24 hour
  energy intake (kcals)

CONTACTS AND LOCATIONS:
Overall Officials: Jill Kanaley, PhD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Misouri, Columbia, Missouri, United States